CLINICAL TRIAL: NCT03570463
Title: GLA:D® Back: Implementation of Group-based Patient Education and Exercises to Support Self-management of Back Pain
Brief Title: GLA:D® Back: Patient Education and Exercises for Self-management of Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Alice Kongsted, Professor wsr, University of Southern Denmark
Other Study IDs: DPA 2015-57-0008 SDU 17/30591
Record Dates: First submitted 2018-05-31; First posted 2018-06-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Back Pain, Low
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GLA:D Back: Two 1-hour group sessions of patient education 8 weeks of twice-weekly 1-hour supervised group exercise sessions
  Interventions: Behavioral: GLA:D Back

INTERVENTIONS:
Behavioral: GLA:D Back — The intervention aims at improving the participant's ability to self-manage low back pain (LBP). The content is based on a cognitive behavioural approach aimed at supporting pain self-efficacy. An individual session at the beginning and the end of the group sessions involve goal-setting and physical tests. Key messages of the patient education include that pain is not a sign of danger and back pain is explained using a behavioural model of (im)balance between demands and capacity rather than emphasising tissue damage. The exercises aim at restoring natural variation in movement and provides guidance for patients in exploring movement rather than teaching exercises in only one correct manner.

SUMMARY:
The GLA:D Back project evaluates the implementation of standardised patient education and exercise therapy for people with persistent or recurrent low back pain (LBP) in a hybrid implementation-effectiveness design. This involves evaluating the process of implementation as well as clinician level outcomes and patient level outcomes.

GLA:D (Good Life with OsteoArthritis in Denmark) is a non-profit initiative and registered trademark from the University of Southern Denmark. It educates clinicians in delivering evidence-based care for musculoskeletal health conditions and registers outcomes in a clinical registry. GLA:D Back uses only the acronym.

The main activity of the implementation strategy is a two-days course for physiotherapists and chiropractors in delivering patient education and exercise therapy that is aimed at supporting patient self-management of LBP. This comes with ready-to-use patient education materials and exercise programs. The course is targeted at chiropractors and physiotherapists, but any health care provider authorised to treat patients with back pain in Denmark can participate, i.e. medical doctors, physiotherapists and chiropractors.

The clinical intervention is a group-based program consisting of two sessions of patient education and 8 weeks of supervised exercises. The program uses a cognitive-behavioural approach and the aim of the exercise component is to restore the patient's ability and confidence to move freely. Clinicians decide which patients are offered the program.

The implementation process is evaluated in a dynamic process monitoring the penetration, adoption and fidelity of the clinical intervention.

The education of clinicians is evaluated via clinician-level outcomes concerning attitudes towards back pain and confidence in managing people with LBP.

The clinical intervention and potential effect mechanisms are evaluated at the patient-level in an observational design. Patients who are participating in the GLA:D Back program are followed using measures of knowledge, skills, beliefs, performance, self-efficacy and success in self-management.

Effects at a national level will be investigated via data from national registries of health care utilisation and sick-leave. Patient- and clinician reported data are collected in a registry.

DETAILED DESCRIPTION:
The clinician training courses are open to all interested authorised back pain clinicians practicing in Denmark. The study evaluates courses conducted in 2018 which involves one or two courses for clinicians in each of five Danish regions.

The adoption of GLA:D Back is investigated by measuring the extent to which clinicians who have participated in the GLA:D Back course conduct the program in their clinics. Reach of the patient target group is determined by asking clinicians about the degree to which patients offered the treatment accept this. Fidelity with the program is investigated quantitatively by asking about treatment content and recall of key messages via patient questionnaires, and by ensuring that patients' individual goals are registered. The quality of care in terms of delivering the key elements of the intervention will be further explored qualitatively.

The profile of patients enrolled in the GLA:D Back programme will be compared between clinics and administrative regions.

Clinician level effects are investigated in an observational longitudinal design with clinician reported data collected before the clinician training course, immediately after the course and 4 months later, and with patient-reported information on delivery collected at their three-months follow up. Indicators of implementation are registration of patients in the GLA:D Back registry and that patients report receiving the educational components of care and supervised exercises. Orientation towards treatment of LBP and confidence in managing patients with LBP are evaluated by clinicians' answers to standardised questionnaires.

Patient level outcomes are aimed at investigating changes in knowledge, beliefs and skills related to the LBP condition which is hypothesized to lead to improved self-efficacy. The initial measures are related to knowledge skills, beliefs and performance, the next line of outcomes to self-efficacy, then daily activities and quality of life and last health care utilisation and work ability.

The compliance with the program is evaluated by patient report of the number of patient education sessions and exercise sessions attended.

The registry is delivered by Odense Patient data Explorative Network (OPEN) at University of Southern Denmark and uses REDCap (Vanderbilt University) as the platform for data collection. Clinicians are registered when signing up for the GLA:D Back course and agreeing to participate in research. Patients are registered by the clinician and have links to patient questionnaires sent to their email before beginning the GLA:D Back program and after 3, 6 and 12 months if consenting to their data being used for research.

Rather than testing effects on one primary outcome, the study evaluates the implementation process and a number of outcomes based on a logical model of change.

ELIGIBILITY:
Inclusion Criteria:

The decision to invite a patient to participate in the GLA:D Back program is at the discretion of the clinician. Clinicians are taught that the program was developed for people with persistent or recurrent low back pain and a need for improved self-management

Exclusion Criteria:

Back pain related to specific spinal or systemic pathology, signs of acute nerve root involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are people consulting a physiotherapist or chiropractor who are trained in the GLA:D Back program. The decision to enrol a patient in GLA:D Back is at the discretion of the clinician in a dialogue with the patient, when clinicians judge that the patient would benefit from improved self-management skills
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Brief Illness Perceptions Questionnaire (B-IPQ) | Change from baseline to 3 months
  Nine items covering the constructs of consequences, timeline (expectations of prognosis), personal control, treatment control, identity (extent of symptoms), coherence (understanding of symptoms), emotional representation, concerns, and cause. Each of the items 1 to 8 are scored 0 - 10. If internal consistency allows so a sum score is calculated (0-80). Cause is registered as text.
Fear Avoidance Beliefs Questionnaire (FABQ) | Change from baseline to 3 months
  FABQ physical activity subscale (0 = no fear avoidance beliefs; 24 = highest possible fear avoidance)
The Arthritis Self-efficacy (ASES) | Change from baseline to 6 months
  ASES subscales of pain and other symptoms. Each item is scored on a 0 - 10 scale (0 = very uncertain; 10 = very certain)
Quality of Life (General health) | Proportions in response categories baseline to 12 months
  The 36-Item Short Form Health Survey (SF-36 item1); 5-point likert scale
Quality of Life (Social functioning) | Change from baseline to 12 months
  The 36-Item Short Form Health Survey (SF-36) subdomain social functioning, transformed score 0-100
Quality of Life (Mental functioning) | Change from baseline to 12 months
  The 36-Item Short Form Health Survey (SF-36) subdomain mental functioning, transformed score 0-100
General Health | Change from baseline to 12 months
  Health thermometer from Eq-5D, score 0= worst imaginable to 100= best imaginable
Health care visits primary care | During 12 months after participation
  Number of primary care visits from national registries
Health care visits hospital | During 12 months after participation
  Number of hospital visits due to LBP from national registries
Imaging | During 12 months after participation
  x-rays, MRI and CT-scans of lower back from national registries
Pain medication | During 12 months after participation
  Prescriptions of pain medication from national registries

SECONDARY OUTCOMES:
Confidence with exercises | Change from baseline to 3 months
  How confident are you in performing exercises in a beneficial way?' (0-10 scale from 'not confident at all' to 'absolutely confident')
Self-assessed physical capacity | Change from baseline to 3 months
  Self-assessed physical fitness visual analogue scales on perceived strength, endurance, flexibility, balance, and moving unhindered as compared with that of other people of the same age and sex. Each item is scored on a 9-point scale (1 = poor; 5 = average; 9 = super). Each item is treated as one subscale
Satisfaction with care | 3 months
  Overall satisfaction with care (5-point Likert scale; 0 = Not at all satisfied, 5 = Extremely satisfied)
Patient reported harms or side effects | 3 months
  Text description of any side effects or problems experienced in relation to the participation in GLA:D Back.
Oswestry Disability Index | Change from baseline to 3, 6, 12 months
  Ten items, sum score 0 - 50 recalculated to 0-100 (0 = No disability; 100 = Maximum disability)
Pain Intensity | Change from baseline to 3, 6, 12 months
  Numeric Rating Scale 0-10 for typical back pain last week (0 = no pain; 10 = worst imaginable pain)
Work ability | During 12 months after participation
  Number of days off work after 1 month of absenteeism available from the 'DREAM' registry from the Danish Ministry of Employment
Brief Illness Perceptions Questionnaire (B-IPQ) | Change from baseline to 6, 12 months
  Nine items covering the constructs of consequences, timeline (expectations of prognosis), personal control, treatment control, identity (extent of symptoms), coherence (understanding of symptoms), emotional representation, concerns, and cause. Each of the items 1 to 8 are scored 0 - 10. If internal consistency allows so a sum score is calculated (0-80). Cause is registered as text.
Fear Avoidance Beliefs Questionnaire (FABQ) | Change from baseline to 6, 12 months
  FABQ physical activity subscale (0 = no fear avoidance beliefs; 24 = highest possible fear avoidance)
The Arthritis Self-efficacy (ASES) | Change from baseline to 3, 12 months
  ASES subscales of pain and other symptoms. Each item is scored on a 0 - 10 scale (0 = very uncertain; 10 = very certain)
Quality of Life (General Health) | Proportions in response categories baseline to 3, 6 months
  The 36-Item Short Form Health Survey (SF-36 item 1),5-point Likert scale
Quality of Life (Social functioning) | Change from baseline to 3, 6 months
  The 36-Item Short Form Health Survey (SF-36) subdomains social functioning, transformed score 0-100
Quality of Life /Mental functioning) | Change from baseline to 3, 6 months
  The 36-Item Short Form Health Survey (SF-36) subdomains of mental functioning, transformed score 0-100

OTHER OUTCOMES:
The Pain Attitudes and Beliefs Scale for Physiotherapists (PABS-PT) | Change from before course participation to 4 months
  Clinician reported 19-item scale. Two subscales: biomedical orientation and behavioural orientation are scored
Practitioner Confidence Scale (PCS) | Change from before course participation to 4 months
  Clinician reported 4-item scale plus two items added to capture confidence about using a behavioral pain model
The Determinants of Implementation Behavior Questionnaire (DIBQ) | Immediately after curse participation and 4 months
  Clinician level measure of the implementation process. Thirty-one items from the domains of knowledge, skills, beliefs about capability, beliefs about consequences, innovation, patients, intentions, organisation, social influences, social context, behavioural regulation, and innovation strategy
Adoption | Within 6 months
  Proportion of clinicians participating in a GLA:D Back course that delivers the program
Patients participation | 4 months
  Clinician reported proportion of invited patients who decide to participate
Patient compliance | 3 months
  Proportion of patients enrolled in GLA:D Back that complete the program

CONTACTS AND LOCATIONS:
Overall Officials: Alice Kongsted, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark (central unit), Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kjaer P, Kongsted A, Ris I, Abbott A, Rasmussen CDN, Roos EM, Skou ST, Andersen TE, Hartvigsen J. GLA:D(R) Back group-based patient education integrated with exercises to support self-management of back pain - development, theories and scientific evidence. BMC Musculoskelet Disord. 2018 Nov 29;19(1):418. doi: 10.1186/s12891-018-2334-x. PMID 30497440
- [Background] Kongsted A, Hartvigsen J, Boyle E, Ris I, Kjaer P, Thomassen L, Vach W. GLA:D(R) Back: group-based patient education integrated with exercises to support self-management of persistent back pain - feasibility of implementing standardised care by a course for clinicians. Pilot Feasibility Stud. 2019 May 9;5:65. doi: 10.1186/s40814-019-0448-z. eCollection 2019. PMID 31086676
- [Background] Kongsted A, Ris I, Kjaer P, Vach W, Morso L, Hartvigsen J. GLA:D(R) Back: implementation of group-based patient education integrated with exercises to support self-management of back pain - protocol for a hybrid effectiveness-implementation study. BMC Musculoskelet Disord. 2019 Feb 18;20(1):85. doi: 10.1186/s12891-019-2443-1. PMID 30777049
- [Background] Ris I, Boyle E, Myburgh C, Hartvigsen J, Thomassen L, Kongsted A. Factors influencing implementation of the GLA:D Back, an educational/exercise intervention for low back pain: a mixed-methods study. JBI Evid Implement. 2021 May 10;19(4):394-408. doi: 10.1097/XEB.0000000000000284. PMID 33965996
- [Background] Morso L, Bogh SB, Ris I, Kongsted A. Mind the gap - Evaluation of the promotion initiatives for implementation of the GLA:D(R) back clinician courses. Musculoskelet Sci Pract. 2021 Jun;53:102373. doi: 10.1016/j.msksp.2021.102373. Epub 2021 Mar 27. PMID 33823485
- [Background] Ris I, Broholm D, Hartvigsen J, Andersen TE, Kongsted A. Adherence and characteristics of participants enrolled in a standardised programme of patient education and exercises for low back pain, GLA:D(R) Back - a prospective observational study. BMC Musculoskelet Disord. 2021 May 22;22(1):473. doi: 10.1186/s12891-021-04329-y. PMID 34022826
- [Background] Joern L, Kongsted A, Thomassen L, Hartvigsen J, Ravn S. Pain cognitions and impact of low back pain after participation in a self-management program: a qualitative study. Chiropr Man Therap. 2022 Feb 21;30(1):8. doi: 10.1186/s12998-022-00416-6. PMID 35189908
- [Background] Nim CG, Kongsted A, Downie A, Vach W. Temporal stability of self-reported visual back pain trajectories. Pain. 2022 Nov 1;163(11):e1104-e1114. doi: 10.1097/j.pain.0000000000002661. Epub 2022 Apr 25. PMID 35467586
- See also: Odense Patient data Explorative Network — https://open.rsyd.dk/OpenProjects/openProject.jsp?openNo=454&lang=da
- See also: Project website — http://gladryg.sdu.dk/
- See also: Data management plan — https://dmp.deic.dk/plans/1737/export.pdf?export%5Bquestion_headings%5D=true